CLINICAL TRIAL: NCT01266759
Title: Combined Contraceptive Vaginal Ring or Norethisterone for Treatment of Idiopathic Menorrhagia
Brief Title: Efficacy of Combined Contraceptive Vaginal Ring(NuvaRing)in Women With Idiopathic Menorrhagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Dr. Hatem Abu Hashim, Associate Prof. of OB/GYN, Mansoura Faculty of Medicine, Mansoura University.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-261z; FMH-245-C
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Menorrhagia
Keywords: Menorrhagia; Vaginal ring; Norethisterone Acetate
MeSH Terms: conditions — Menorrhagia | interventions — NuvaRing; Norethindrone Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NuvaRing (Experimental): For the first cycle, women inserted the ring between days 1 and 5 of the menstrual cycle. Treatment continued for three cycles. Each cycle consisted of 3 weeks of ring use followed by a 1 week ring-free period.
  Interventions: Drug: NuvaRing
- Norethisterone Acetate (Active Comparator): Norethisterone Acetate tablets at a dose of 5 mg three times daily from day 5 to 26 of the cycle over three cycles. Male condom used for contraception during treatment
  Interventions: Drug: Norethisterone Acetate tablets - 5mg

INTERVENTIONS:
Drug: NuvaRing — For the first cycle, women inserted the ring between days 1 and 5 of the menstrual cycle. Treatment continued for three cycles. Each cycle consisted of 3 weeks of ring use followed by a 1 week ring-free period.
  Arms: NuvaRing
Drug: Norethisterone Acetate tablets - 5mg — Norethisterone Acetate tablets 5 mg three times daily from day 5 to 26 of the cycle over three cycles. Male condom used for contraception during treatment
  Arms: Norethisterone Acetate

SUMMARY:
To compare the efficacy of a combined contraceptive vaginal ring (NuvaRing) and oral Norethisterone Acetate in treatment of Idiopathic heavy menstrual bleeding during fertile age

ELIGIBILITY:
Inclusion Criteria:

* Women with heavy menstrual bleeding based on PBAC score over 185 (mean of two control cycles)and desire contraception

Exclusion Criteria:

* Menorrhagia of endocrine or systemic origin
* other pathology e.g. patients with fibroids of any size, adenomyosis, endometriosis, pelvic inflammatory disease.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2008-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Reduction in menstrual blood loss at the end of study (cycle 3) measured by pictorial blood loss assessment chart.

SECONDARY OUTCOMES:
Haemoglobin and serum ferritin at the end of study (cycle 3)

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD MRCOG, Principal Investigator — Mansoura University Hospital; Waleed El-Sherbini, MD, Study Director — Mansoura University Hospital; Mohamed Bazeed, MD, Study Chair — Mansoura University Hospital
Locations (1):
- Mansoura University Hospitals,OB/GYN department, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Matteson KA, Boardman LA, Munro MG, Clark MA. Abnormal uterine bleeding: a review of patient-based outcome measures. Fertil Steril. 2009 Jul;92(1):205-16. doi: 10.1016/j.fertnstert.2008.04.023. Epub 2008 Jul 16. PMID 18635169
- [Background] Oddsson K, Leifels-Fischer B, Wiel-Masson D, de Melo NR, Benedetto C, Verhoeven CH, Dieben TO. Superior cycle control with a contraceptive vaginal ring compared with an oral contraceptive containing 30 microg ethinylestradiol and 150 microg levonorgestrel: a randomized trial. Hum Reprod. 2005 Feb;20(2):557-62. doi: 10.1093/humrep/deh604. Epub 2004 Nov 11. PMID 15539438